CLINICAL TRIAL: NCT03682497
Title: A Phase I, Open Label, Randomized, Parallel Group, Multicentre Study to Compare the Effect of AZD9977 and Spironolactone on Serum Potassium [sK+] During 28 Days in Patients With HFmrEF or HFpEF and eGFR in the Range of ≥40 and ≤70 mL/Min/1.73m2.
Brief Title: Study in HFpEF Patients to Compare the Effect of AZD9977 and Spironolactone on Serum Potassium
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Attendance at study sites carries risk of COVID-19 infection. Non-attendance at planned study site visits has unacceptable study related patient safety risk.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6401C00004
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure
Keywords: Heart failure.; Oral selective mineralocorticoid receptor modulator.; Heart failure with preserved ejection fraction (HFpEF).
MeSH Terms: conditions — Heart Failure | interventions — AZD9977; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spironolactone (Active Comparator): Spironolactone treatment for 28 days
  Interventions: Drug: Spironolactone
- AZD9977 (Experimental): AZD9977 treatment for 28 days
  Interventions: Drug: AZD9977

INTERVENTIONS:
Drug: AZD9977 — AZD9977 capsules taken orally for 28 days.
  Arms: AZD9977
Drug: Spironolactone — Spironolactone tablets taken orally for 28 days.
  Arms: Spironolactone

SUMMARY:
This is a Phase I, Multicentre study to Compare the Effect of AZD9977 and Spironolactone on Serum Potassium [sK+] during 28 days in Patients with HFmrEF or HFpEF and eGFR in the range of ≥40 and ≤70 mL/min/1.73m2.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and signs consistent with a diagnosis of heart failure (HF)
* Left ventricular ejection fraction (LVEF) ≥40% by transthoracic echocardiography within the past 12 months
* Plasma NT-proBNP level ≥125 pg/ml (≥ 600pg/mL if patient has persistent or permanent atrial fibrillation, atrial flutter, or atrial tachycardia)
* Estimated glomerular filtration rate (eGFR) ≥40 and ≤70ml/min/1.73m2 (by CKD-EPI formula).
* Baseline serum potassium (sK+) level ≥3.5 and ≤4.8mmol/l.
* Stable doses of the following medications at baseline for at least 4 weeks prior to randomisation:

Angiotensin receptor blocker (ARB) or Angiotensin converting enzyme inhibitor (ACEi) Loop diuretic (up to a 120mg furosemide dose or equivalent

Exclusion Criteria:

* Patients with documented LVEF <40% at any time (i.e. patients with previously impaired LVEF that has now improved are not permitted).
* Patients experiencing acute decompensation of heart failure requiring hospital admission or escalation in therapy.
* Primary cardiomyopathy (e.g. constrictive, restrictive, infiltrative, toxic, hypertrophic, congenital or any primary cardiomyopathy in judgment of Investigator).
* Hyponatraemia, defined as serum Na+ <135 mmol/L at the time of enrollment.
* Persistent resting sinus tachycardia >110 bpm or sinus bradycardia <45bpm.
* Systolic blood pressure (BP) <110mmHg or >180mmHg.
* Diastolic BP <60 mmHg or >100 mmHg.
* Patients previously intolerant to MRA (e.g. spironolactone or eplerenone) for any reason.
* Medical conditions associated with development of hyperkalaemia (e.g. Addison's disease).
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥2.0 times the upper limit of normal (ULN).
* Patients who have been taking an MR antagonist within 1 month prior to randomization.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Relative change (%) from baseline in serum potassium | Measurements on day 1, 7, 14, 21 and 28 will be used. The primary comparison between Spironolactone and AZD9977 will be done at day 28.
  To compare the effect of AZD9977 with spironolactone on serum potassium (sK+)

SECONDARY OUTCOMES:
Plasma trough concentrations (Ctrough) values of spironolactone and AZD9977 | PK samples will be taken (within 60 min prior to dose) at day 1, 7, 14, 21 and 28.
  To evaluate the pharmacokinetics (PK) of AZD9977 and spironolactone
Relative change (%) from baseline in serum potassium | Measurements on day 1, 7 and 14 will be used. The primary comparison between Spironolactone and AZD9977 will be done at day 14.
  To compare the effects of AZD9977 with spironolactone on serum potassium at Day 14.

CONTACTS AND LOCATIONS:
Locations (16):
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Czechia (6):
  - Research Site, Brandýs nad Labem
  - Research Site, Česká Lípa
  - Research Site, Jaroměř
  - Research Site, Louny
  - Research Site, Pardubice
  - Research Site, Prague
- Poland (5):
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Legnica
  - Research Site, Warsaw
  - Research Site, Wroclaw
- United Kingdom (3):
  - Research Site, Hull
  - Research Site, Leicester
  - Research Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home